CLINICAL TRIAL: NCT04551287
Title: Artificial Intelligence Enables Precision Diagnosis of Cervical Cytology Grades and Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: 2020-KY-114
Record Dates: First submitted 2020-09-06; First posted 2020-09-16 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Cervical Cancer; Diagnostic Platform; Diagnosing Cervical Cytology Grades and Cancer; Artificial Intelligence
Keywords: Diagnostic Platform; Cervical Cytology Grade Diagnosis; Thinprep Cytologic Test; Artificial Intelligence Deep Learning Algorithm
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Samples Without DNA: Samples retained, with no potential for DNA extraction from any retained samples (e.g., fixed tissue, plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Training dataset: 11,468 eligible individuals' slides for the cervical cytology screening collected from the Sun Yat-sen Memorial Hospital (SYSMH, Guangzhou, China) between January 2016 and January 2020, were randomly assigned to the training dataset (n = 9,316) and the internal validation dataset (n = 2,152) in order to train and validate the Artificial Intelligence Cervical Cancer Screening (AICS).
- SYSMH internal validation dataset: 11,468 eligible individuals' slides for the cervical cytology screening collected from the Sun Yat-sen Memorial Hospital (SYSMH, Guangzhou, China) between January 2016 and January 2020, were randomly assigned to the training dataset (n = 9,316) and the internal validation dataset (n = 2,152) in order to train and validate the Artificial Intelligence Cervical Cancer Screening (AICS).
- TAHGMU external validation dataset: 600 slides from 600 eligible individuals were obtained in the Third Affiliated Hospital of Guangzhou Medical University (TAHGMU, Guangzhou, China) between January 2016 and January 2020, which was used to validate the Artificial Intelligence Cervical Cancer Screening (AICS).
- GWCMC external validation dataset: 600 slides from 600 eligible individuals were obtained in Guangzhou Women and Children Medical Center (GWCMC, Guangzhou, China) between January 2016 and January 2020, which was used to validate the Artificial Intelligence Cervical Cancer Screening (AICS).
- Prospective validation dataset: A prospective validation dataset was conducted to distinguish the diagnostic performance of the cytopathologists, AICS, and AICS-assisted cytopathologists, in which 2,780 eligible slides from 2,780 individuals were obtained and prospectively labeled between August 28, 2020 and October 16, 2020 at SYSMH.
- Randomized controlled trial: A prospective randomized controlled trial was conducted to compare the performance of the cytopathologists, AICS, and AICS-assisted cytopathologists in SYSMH. Here, 618 slides were collected between August 13, 2020, and December 14, 2020, to build the SYSMH randomized controlled trial. The remaining 608 slides after quality control were randomly assigned (1:1:1) to the AICS group (n = 201), the cytopathologists group (n = 203), and the AICS-assisted cytopathologists group (n = 204).

SUMMARY:
Cervical cancer, the fourth most common cancer globally and the fourth leading cause of cancer-related deaths, can be effectively prevented through early screening. Detecting precancerous cervical lesions and halting their progression in a timely manner is crucial. However, accurate screening platforms for early detection of cervical cancer are needed. Therefore, it is urgent to develop an Artificial Intelligence Cervical Cancer Screening (AICS) system for diagnosing cervical cytology grades and cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women Aged 25-65 years old.
2. Availability of confirmed diagnostic results of the cervical liquid-based cytological examination, and satisfactory digital images from the liquid-based cytology pap test: at least 5000 uncovered and observable squamous epithelial cells, samples with abnormal cells (atypical squamous cells or atypical glandular cells and above).

Exclusion Criteria:

1. Unsatisfactory samples of cervical liquid-based cytological examination: less than 5000 uncovered, observable squamous epithelial cells, and more than 75% of squamous epithelial cells affected because of blood, inflammatory cells, epithelial cells over-overlapping, poor fixation, excessive drying, or contamination of unknown components.
2. Women diagnosed with other malignant tumors other than cervical cancer.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients who were 18 years or older with clear diagnostic results of cervical liquid-based cytological examination were included. All cases were collected from Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University.
Sampling Method: Non-Probability Sample
Enrollment: 16164 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Area under ROC curve (AUC) | Diagnostic evaluation will be performed within 1 week when the smear pictures are obtained
  Area under the curve

SECONDARY OUTCOMES:
Specificity | Diagnostic evaluation will be performed within 1 week when the smear pictures are obtained
  The true negative rate (TNR) of the diagnostic platform, which is the ratio between the number of negative individuals correctly categorized by platform and the total number of actual negative individuals (%).
Sensitivity | Diagnostic evaluation will be performed within 1 week when the smear pictures are obtained
  The true positive rate (TPR) of the diagnostic platform, which is the ratio between the number of positive individuals correctly categorized by platform and the total number of actual positive individuals (%).
Accuracy | Diagnostic evaluation will be performed within 1 week when the smear pictures are obtained
  The quantity of true positive (TP) plus true negative (TN) over the quantity of (TP) plus true negative (TN) plus false positive (FP) plus false negative (FN).

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (3):
- China (3):
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No
Requests for the data collected and analyzed in this study will be considered if the application is in line with public benefits and the applicant is willing to sign a data access agreement. Contact can be through the corresponding author.